CLINICAL TRIAL: NCT05844358
Title: PROSPECTIVE MULTICENTRIC CLINICAL STUDY TO ASSESS SAFETY OF A CORTICAL BONE TRAJECTORY SCREW INSERTION TECHNIQUE WITH THE USE OF PATIENT SPECIFIC DRILL GUIDES
Brief Title: Cortical Bone Trajectory With Patient Guide
Acronym: MySpine MC
Status: Completed | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P05.007.05
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: MySpine MC — Spinal stabilization throught the support of patient specific guide, MySpine MC according to cortical bone trajectory technique

SUMMARY:
The use of patient specific guides with proper preoperative planning, following a cortical bone trajectory technique, should guarantee a successful surgery and benefit of less invasive technique.

This study intends to measure the safety and efficacity of MySpine MC patient-specific guide system, when used according to its general indication of use and following the surgical technique suggested by the manufacturer

DETAILED DESCRIPTION:
Adult patients affected by degenerative disc disease, meeting all inclusion/exclusion criteria, will be proposed to take part to the current post-marketing surveillance study during their pre-operative visit. They will be provided with an information letter and, in case of acceptance to participate to the study, asked to sign a consent form.

After enrolment, each patient will be monitored for 13 months. Data concerning demography, preoperative clinical conditions, surgical details including device implanted and complications occurred, postoperative clinical and/or radiological assessments (as per standard routine at 5 weeks, 3, 7 and 13 months) will be prospectively collected. The level of bone fusion will be evaluated with a postoperative CT scan at 7 ±2 months follow-up

ELIGIBILITY:
Inclusion Criteria:

1. those affected by degenerative disc disease needing a surgical treatment one/two levels with posterior approach to screw fixation
2. those who need a surgical procedure of lumbar spine stabilization according to Medacta device instruction for use from level L2 to level S1
3. those who signed consent form to participate to the study
4. Normal healthy patients or with mild systematic disease identified as patients with ASA score 1 or 2
5. Patients with BMI ≤ 35 kg/m2
6. non responsive or unsufficient resposive to non -invasive treatment such as analgesics

Exclusion Criteria:

1. Patients affected by lytic lystesis and degenerative lystesis with grade≥2 will be excluded
2. Patients <18 years
3. Patient who is pregnant or intends to become pregnant during the study
4. Known substance or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A consecutive ongoing recruitment through study members in daily clinical practice will take place.
  The 102 patients planned for this survey will be recruited by the Investigators meeting all the inclusion/exclusion criteria.
  Subjects, among those whose clinical condition makes them eligible for a spinal stabilization, will be invited to participate to the study. Enrolment will take place over a period of 24 months, until the forecasted number of 102 patients has entered into the survey.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Bone fusion | 6 months
  Percentage of subjects get bone fusion at index level will be calculated

SECONDARY OUTCOMES:
Pain perception | preop, 5 weeks, 3months, 6 months, 12 months
  A visual analog scale will be filled to assess leg and back pain
Functional status | preop, 5 weeks, 3months, 6 months, 12 months
  ODI index questionnaire for assessing functional status and quality-of-life impairment in patients with low back pain or spinal cord disease and injury in research and clinical settings will be filled
Quality of life | preop, 5 weeks, 3months, 6 months, 12 months
  Euroqol 5D questionnaire will be collected to assess quality of life
Safety device | preop, 5 weeks, 3months, 6 months, 12 months
  collection of adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Geert Mahieu, Dr, Principal Investigator — AZ Monica Hospital; Patricia Verstraete, Dr, Principal Investigator — AZ Sint-Elisabeth Turnhout
Locations (2):
- Belgium (2):
  - AZ Monica Hospital, Antwerp
  - AZ Sint-Elisabeth Turnhout, Turnhout

IPD SHARING:
Plan to Share IPD: No